CLINICAL TRIAL: NCT04109378
Title: The Impact of NOSE-colectomy on Fertility and Quality of Life Among Patients With Colorectal Endometriosis
Acronym: NOSERES
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Semmelweis University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SemmlweisU
Record Dates: First submitted 2019-08-26; First posted 2019-09-30 (Actual); Last update posted 2022-05-17 (Actual); Status verified 2022-05

CONDITIONS: Endometriosis; Quality of Life
Keywords: Fertility; Colorectal endometriosis; Surgery
MeSH Terms: conditions — Endometriosis

STUDY DESIGN:
Intervention Model Description: Our study was designed as a two-arm prospective randomized trial where all cases will be executed unblindly. As an experimental clinical trial the cases have been managed independently where the applied measures were computer based randomization.
  In addition clustering effect has been examined within the two groups. The statistical power will be calculated for a sample size.
  Randomization: Blinding in our study is not feasible.
  Assignment of a patient to conventional or NOSE-colorectal resection is based on a randomization list using the simple randomization method. In order to determine the allocation sequence a computer based (www.random.org) coin flipping is carried out by a staff member with no clinical involvement in the study. The randomization will start after the patient had completed all baseline assessments and had given written consent to be enrolled in the trial.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients operated with conventional laparoscopic technique (Active Comparator): Patients operated with conventional laparoscopic technique for colorectal DIE
  Interventions: Procedure: Surgical procedures( conventional laparoscopic and NOSE technique) for the treatment of colorectal DIE
- Patients operated with NOSE laparoscopic technique (Active Comparator): Patients operated with NOSE technique for colorectal DIE
  Interventions: Procedure: Surgical procedures( conventional laparoscopic and NOSE technique) for the treatment of colorectal DIE

INTERVENTIONS:
Procedure: Surgical procedures( conventional laparoscopic and NOSE technique) for the treatment of colorectal DIE — For conventional laparoscopic and NOSE techniques a 4-port approach is used. The rectum is skeletonized. The distal rectum is closed using an endoscopic linear stapler. The mobilized rectum with the specimen is retrieved through a small suprapubic incision. The anvil of a conventional circular stapler is introduced in the proximal colon after placement of a purse string suture. A circular stapled colorectal anastomosis is fired. In case of NOSE, both the proximal sigmoid colon and the proximal rectum are tied off laparoscopically with a nonabsorbable suture. A transverse colotomy is performed in healthy tissue using a harmonic scalpel to deliver the anvil from a circular stapler introduced through the anus. The specimen is extracted transrectally in a specimen retrieval bag. Proximal part of the anastomosis is completed by suturing the anvil in place with a laparoscopic suture. The distal rectum is closed using a linear stapler. End-to-end anastomosis is made using the circular stapler

SUMMARY:
Deep infiltrating endometriosis (DIE) represents the most severe form of endometriosis and is present in 20-35% of all women suffering from the disease. Intestinal nodules are observed in 3% to 37% of endometriosis patients. In cases of colorectal DIE, adequate therapy depends on the depth of infiltration and the size of the lesion as well as the woman's quality of life. Removal of the specimen after segmental bowel resection can be performed by either mini-laparotomy or by the natural orifice specimen extraction (NOSE) technique .

The assessment of the quality of life and fertility outcome of the patients was done by using electronic questionnaires before and after surgery.

DETAILED DESCRIPTION:
Endometriosis is an enigmatic disease affecting 6-10% of women of reproductive age or 176 millions of women worldwide (1). Endometriosis is defined as the presence of endometrial-like tissue outside the uterus and it induces a chronic inflammatory reaction (2). Deep infiltrating endometriosis (DIE) represents the most severe form of endometriosis (described by the invasion of anatomical structures and organs deeper than 5 mm beyond the peritoneum) and is present in 20-35% of all women suffering from the disease (3). Intestinal deep infiltrating endometriosis is known as lesions infiltrating at least the muscular layer of the bowel wall and most commonly affects the rectum, sigmoid colon and the rectovaginal septum. (4).

Even if bowel endometriosis may be totally asymptomatic, in many patients intestinal wall DIE alters significantly quality of life by provoking constipation, diarrhea, hematochezia, intestinal cramping, abdominal bloating, intestinal stenosis or obstruction and pain of defecation (5, 6). Rectal fixation to adjacent structures results in angulation of the rectum and subsequent defecatory pain and constipation. Fibrosis of nodules can lead to rectal constriction and stenosis, cyclical inflammation of the rectal wall may lead to changes in bowel habit (usually diarrhoea) with or without rectal bleeding (7).

Although the surgical laparoscopic management of endometriosis is widely accepted, the optimal type of resection, whether conservative approach (shaving, disc resection) or radical technique (involves limited resection of the bowel wall with preservation of all adjacent structures-autonomic pelvic plexus, rectal vascular supply- known as "nerve-vessel sparing limited segmental resection"), is under discussion for treatment of deep endometriosis infiltrating the rectum.

In cases of colorectal DIE, adequate therapy depends on the precise location, extent of the nodule and depth of invasion, as well as the woman's quality of life (3). Removal of the specimen after segmental bowel resection can be performed by either mini-laparotomy (conventional method) or by the natural orifice specimen extraction (NOSE) technique. (8).

The conventional method raises concerns because this could disrupt the integrity of the abdominal wall. Moreover, extraction site laparotomy is associated with higher postoperative pain scores. The occurrence of particular complications such as incisional hernias and wound infections is also higher than after conventional laparoscopic procedures (8).

In order to avoid these complications, NOSE technique has been introduced. During NOSE colectomy the specimen is extracted through a natural orifice and an intracorporeal anastomosis is performed (8).

Several studies have demonstrated a significant drop in pain scores and amelioration of impaired sexual functioning and improved pregnancy rates in women following surgical resection of colorectal endometriosis (9).

The aim of this study is to report the short, medium and long-term bowel functional outcomes and improvement of infertility, quality of life in women undergoing conventional and NOSE segmental bowel resection for endometriosis at our institution using validated questionnaires.

Functional and psychological outcomes will be assessed using different questionnaires at baseline and postoperative follow-up moments.

* Endometriosis Health Profile, EHP 30 (10)
* Gastrointestinal Quality of Life Index, GIQLI (11)
* Low Anterior Resection Syndrome score, LARS (12)
* Assessment of endometriosis related pain: Visual Analog Scale (13)
* Psychological questionnaires: Pain catastrophizing Scale (14), Self-Efficacy for Managing Chronic Disease 6-item Scale (15).

ELIGIBILITY:
Inclusion criteria:

* Age: 18 - 45 years (both inclusive)
* Complaining of infertility and/or pain
* Deep endometriosis infiltrating the rectum on at least one imaging technique or confirmed by previous surgery

  * up to 15 cm from the anus
  * Involving at least the muscularis layer in depth

Exclusion criteria

A potential subject who meets any of the following criteria will be excluded from participation in this study:

* Suspected pelvic malignancy
* Pregnancy
* Patients without bowel resection

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Hundred and fifty (n=150) premenopausal women with deep infiltrating endometriosis of the rectum who are scheduled for surgical treatment for DIE in our institution during the time will be included in the study.
  All women with suspicion of a deep endometriosis will be examined (gynecological examination) by a surgeon experienced in endometriosis. For further mapping of the endometriosis following imaging techniques will be used:
  * Transvaginal ultrasound using the IDEA terminology to describe the endometriotic lesions found (17)
  * Complementary examinations can be needed depending on the lesions that are found. For example, MR examination, or intravenous pyelogram in women with associated involvement of the urine tract.
Enrollment: 150 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2021-03-23 (Actual); Study Completion 2021-03-23 (Actual)

PRIMARY OUTCOMES:
Endometriosis Health Profile, EHP 30 | 24 months
  To describe the difference in patient reported outcomes after conventional segmental bowel resection treatment in comparison to NOSE colectomy in patients with deep endometriosis infiltrating the rectum.
  The patients are asked to fill the questionnaires preoperatively, at 30 days, 6 months, 1 year and 2 years after the surgery. During the present study investigators are planning an average follow-up of 24 months.
  Impact of surgical technique on the quality of life. The outcome will be assessed using validated electronic questionnaires containing questions from Endometriosis Health Profile 30. This is a core questionnaire which consists of five scales (pain, control and powerlessness, emotional well-being, social support, and self-image) contains a total of 30 items. (10)
Gastrointestinal Quality of Life Index, GIQLI | 24 months
  To describe the difference in patient reported outcomes after conventional segmental bowel resection treatment in comparison to NOSE colectomy in patients with deep endometriosis infiltrating the rectum.
  The patients are asked to fill the questionnaires preoperatively, at 30 days, 6 months, 1 year and 2 years after the surgery. During the present study investigators are planning an average follow-up of 24 months.
  GIQLI is a 36-item patient reported outcomes instrument designed to assess GI-specific health-related quality of life in clinical practice of patients with gastrointestinal disorders. It has five domains (GI symptoms, emotion, physical function, social function and medical treatment) and subscores range from 0-4 while the total score range from 0-144. Higher scores mean better GI health-related quality of life. (11)
LARS score before and after colorectal resection for DIE | 24 months
  To describe the difference in patient reported outcomes after conventional segmental bowel resection treatment in comparison to NOSE colectomy in patients with deep endometriosis infiltrating the rectum.
  The patients are asked to fill the questionnaires preoperatively, at 30 days, 6 months, 1 year and 2 years after the surgery. During the present study investigators are planning an average follow-up of 24 months.
  The Low Anterior Resection Syndrome (LARS) is a common complication that occures after colorectal surgery. The LARS score is a simple self-administered questionnaire measuring bowel dysfunction after rectal surgery. Contains questions regarding incontinence, emptying difﬁculties, urgency, and frequency. The calculated score ranges from 0 to 42, with a score of 0-20 representing no LARS, a score of 21-29 representing minor LARS and a score of 30-42 representing major LARS. (12)
Endometriosis related pain before and after colorectal resection for DIE | 24 months
  To describe the difference in patient reported outcomes after conventional segmental bowel resection treatment in comparison to NOSE colectomy in patients with deep endometriosis infiltrating the rectum.
  The patients are asked to fill the questionnaires preoperatively, at 30 days, 6 months, 1 year and 2 years after the surgery. During the present study investigators are planning an average follow-up of 24 months.
  For the assessment of pre- and postoperative pain a Visual Analogue Scale is used (from 1-10, where 1 is the lowest and 10 is the maximum score) to assess the pre- and postoperative quality of life (dysmenorrhoea, dyspareunia, dyschezia, dysuria, CPP) (13).
Infertility outcomes after colorectal resection for bowel endometriosis | 24 months
  Number of pregnancies, cumulative pregnancy rate and take home baby rate after laparoscopic bowel resection.
Psychological questionnaires: | 24 months
  To describe the difference in patient reported outcomes after conventional segmental bowel resection treatment in comparison to NOSE colectomy in patients with deep endometriosis infiltrating the rectum.
  The patients are asked to fill the questionnaires preoperatively, at 30 days, 6 months, 1 year and 2 years after the surgery. During the present study investigators are planning an average follow-up of 24 months.
  Pain catastrophizing Scale, Self-Efficacy for Managing Chronic Disease 6-item Scale to investigate the psychological aspect of the disease (14,15).

SECONDARY OUTCOMES:
Complication rates after conventional and NOSE-colectomy performed for colorectal endometriosis | 24 months
  To measure the complication rates after conventional and NOSE-colectomy performed for colorectal endometriosis. The complication rates between the NOSE vs conventional specimen extraction technique will be examined. The difference between the complication rates will be presented according to Clavien-Dindo Classification System (16).
  As follows:
  Grade I Any deviation from the normal postoperative course without treatment by invasive interventions Grade II Requiring pharmacological treatment with drugs other than such allowed for grade I complications.
  Grade III
  Requiring surgical, endoscopic or radiological intervention
  * IIIa
  Intervention not under general anesthesia
  * IIIb
  Intervention under general anesthesia Grade IV
  Life-threatening complication requiring IC/ICU-management
  * IVa
  single organ dysfunction (including dialysis)
  * IVb
  multiorgan dysfunction Grade V Death of a patient
Hospital stay after colorectal resection perfomed for the treatment of bowel endometriosis | 24 months
  To measure the hospital stay after colorectal resection perfomed for the treatment of bowel endometriosis
Lenght of recovery after colorectal resection performed for the treatment of bowel endometriosis | 24 months
  To measure the lenght of recovery after bowel resection will be assessed by the comparison of the hospital stay (mean +/- SD days)

CONTACTS AND LOCATIONS:
Overall Officials: Attila Bokor, MD, PhD, Study Director — Semmelweis University; Noemi Dobo, MD, Study Chair — Semmelweis University
Locations (1):
- Semmelweis University, Budapest, Hungary

IPD SHARING:
Plan to Share IPD: Yes
Will individual participant data will be available (including datadictionaires)? Individual participant data will be available. What data in particular will be shared? Individual participant data that underline the results reported in the article after deidentification (text, tables, figures and appendices) will be shared.
  What other documents will be available? Study protocol, statistical analysis plan, analytic code will be available as well.
  When will data be available (start and end dates)? Data will be available from 3 months to 5 years after the publication of the article.
  With whom? The data will be shared with researchers who provide a methodologically sound proposal.
  For what types of analysis? To achieve aims in the approved proposal. By what mechanism will data be made available? Proposals should be directed to attila.z.bokor@gmail.com. To gain access, data requestors will need to sign a data access agreement. Data are available for 5 years.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: 5 years after study closure
Access Criteria: Any researcher intersted in the study

REFERENCES:
- [Background] Simoens S, Dunselman G, Dirksen C, Hummelshoj L, Bokor A, Brandes I, Brodszky V, Canis M, Colombo GL, DeLeire T, Falcone T, Graham B, Halis G, Horne A, Kanj O, Kjer JJ, Kristensen J, Lebovic D, Mueller M, Vigano P, Wullschleger M, D'Hooghe T. The burden of endometriosis: costs and quality of life of women with endometriosis and treated in referral centres. Hum Reprod. 2012 May;27(5):1292-9. doi: 10.1093/humrep/des073. Epub 2012 Mar 14. PMID 22422778
- [Background] Kennedy S, Bergqvist A, Chapron C, D'Hooghe T, Dunselman G, Greb R, Hummelshoj L, Prentice A, Saridogan E; ESHRE Special Interest Group for Endometriosis and Endometrium Guideline Development Group. ESHRE guideline for the diagnosis and treatment of endometriosis. Hum Reprod. 2005 Oct;20(10):2698-704. doi: 10.1093/humrep/dei135. Epub 2005 Jun 24. PMID 15980014
- [Background] Wolthuis AM, Tomassetti C. Multidisciplinary laparoscopic treatment for bowel endometriosis. Best Pract Res Clin Gastroenterol. 2014 Feb;28(1):53-67. doi: 10.1016/j.bpg.2013.11.008. Epub 2013 Dec 2. PMID 24485255
- [Background] Meuleman C, Tomassetti C, D'Hoore A, Van Cleynenbreugel B, Penninckx F, Vergote I, D'Hooghe T. Surgical treatment of deeply infiltrating endometriosis with colorectal involvement. Hum Reprod Update. 2011 May-Jun;17(3):311-26. doi: 10.1093/humupd/dmq057. Epub 2011 Jan 13. PMID 21233128
- [Background] Kossi J, Setala M, Makinen J, Harkki P, Luostarinen M. Quality of life and sexual function 1 year after laparoscopic rectosigmoid resection for endometriosis. Colorectal Dis. 2013 Jan;15(1):102-8. doi: 10.1111/j.1463-1318.2012.03111.x. PMID 22642851
- [Background] Roman H, Bubenheim M, Huet E, Bridoux V, Zacharopoulou C, Darai E, Collinet P, Tuech JJ. Conservative surgery versus colorectal resection in deep endometriosis infiltrating the rectum: a randomized trial. Hum Reprod. 2018 Jan 1;33(1):47-57. doi: 10.1093/humrep/dex336. PMID 29194531
- [Background] Ng A, Yang P, Wong S, Vancaillie T, Krishnan S. Medium to long-term gastrointestinal outcomes following disc resection of the rectum for treatment of endometriosis using a validated scoring questionnaire. Aust N Z J Obstet Gynaecol. 2016 Aug;56(4):408-13. doi: 10.1111/ajo.12476. Epub 2016 Jun 14. PMID 27297610
- [Background] Bokor A, Lukovich P, Csibi N, D'Hooghe T, Lebovic D, Brubel R, Rigo J. Natural Orifice Specimen Extraction during Laparoscopic Bowel Resection for Colorectal Endometriosis: Technique and Outcome. J Minim Invasive Gynecol. 2018 Sep-Oct;25(6):1065-1074. doi: 10.1016/j.jmig.2018.02.006. Epub 2018 Feb 14. PMID 29454144
- [Background] Hudelist G, Aas-Eng MK, Birsan T, Berger F, Sevelda U, Kirchner L, Salama M, Dauser B. Pain and fertility outcomes of nerve-sparing, full-thickness disk or segmental bowel resection for deep infiltrating endometriosis-A prospective cohort study. Acta Obstet Gynecol Scand. 2018 Dec;97(12):1438-1446. doi: 10.1111/aogs.13436. Epub 2018 Sep 16. PMID 30080244
- [Background] Jones G, Kennedy S, Barnard A, Wong J, Jenkinson C. Development of an endometriosis quality-of-life instrument: The Endometriosis Health Profile-30. Obstet Gynecol. 2001 Aug;98(2):258-64. doi: 10.1016/s0029-7844(01)01433-8. PMID 11506842
- [Background] Eypasch E, Williams JI, Wood-Dauphinee S, Ure BM, Schmulling C, Neugebauer E, Troidl H. Gastrointestinal Quality of Life Index: development, validation and application of a new instrument. Br J Surg. 1995 Feb;82(2):216-22. doi: 10.1002/bjs.1800820229. PMID 7749697
- [Background] Emmertsen KJ, Laurberg S. Low anterior resection syndrome score: development and validation of a symptom-based scoring system for bowel dysfunction after low anterior resection for rectal cancer. Ann Surg. 2012 May;255(5):922-8. doi: 10.1097/SLA.0b013e31824f1c21. PMID 22504191
- [Background] Bourdel N, Alves J, Pickering G, Ramilo I, Roman H, Canis M. Systematic review of endometriosis pain assessment: how to choose a scale? Hum Reprod Update. 2015 Jan-Feb;21(1):136-52. doi: 10.1093/humupd/dmu046. Epub 2014 Sep 1. PMID 25180023
- [Background] Lorig KR, Sobel DS, Ritter PL, Laurent D, Hobbs M. Effect of a self-management program on patients with chronic disease. Eff Clin Pract. 2001 Nov-Dec;4(6):256-62. PMID 11769298
- [Background] Dindo D, Demartines N, Clavien PA. Classification of surgical complications: a new proposal with evaluation in a cohort of 6336 patients and results of a survey. Ann Surg. 2004 Aug;240(2):205-13. doi: 10.1097/01.sla.0000133083.54934.ae. PMID 15273542
- [Background] Guerriero S, Condous G, van den Bosch T, Valentin L, Leone FP, Van Schoubroeck D, Exacoustos C, Installe AJ, Martins WP, Abrao MS, Hudelist G, Bazot M, Alcazar JL, Goncalves MO, Pascual MA, Ajossa S, Savelli L, Dunham R, Reid S, Menakaya U, Bourne T, Ferrero S, Leon M, Bignardi T, Holland T, Jurkovic D, Benacerraf B, Osuga Y, Somigliana E, Timmerman D. Systematic approach to sonographic evaluation of the pelvis in women with suspected endometriosis, including terms, definitions and measurements: a consensus opinion from the International Deep Endometriosis Analysis (IDEA) group. Ultrasound Obstet Gynecol. 2016 Sep;48(3):318-32. doi: 10.1002/uog.15955. Epub 2016 Jun 28. PMID 27349699
- [Derived] Dobo N, Marki G, Hudelist G, Csibi N, Brubel R, Acs N, Bokor A. Laparoscopic natural orifice specimen extraction colectomy versus conventional laparoscopic colorectal resection in patients with rectal endometriosis: a randomized, controlled trial. Int J Surg. 2023 Dec 1;109(12):4018-4026. doi: 10.1097/JS9.0000000000000728. PMID 37720929